CLINICAL TRIAL: NCT05992233
Title: Is Dual-wavelength Low-level Laser Therapy Effective in Reducing Pain, Swelling and Trismus After Impacted Mandibular Third Molar Extraction?
Brief Title: "Effectiveness of Dual-Wavelength Laser Therapy in Third Molar Extraction Pain, Swelling, and Trismus"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, esengul sen, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-KAEK-078
Record Dates: First submitted 2023-04-19; First posted 2023-08-15 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Molar, Third; Low-level Laser Therapy
Keywords: photobiomodulation,; Impacted third molar; Pain; Edema
MeSH Terms: conditions — Pain; Edema

STUDY DESIGN:
Intervention Model Description: hee primary outcome was postoperative pain, evaluated using the visual analogue scale (VAS) score at Baseline, for 7 days following surgery, postoperative swelling and maximum mouth opening values evaluated at 2nd and 7th days in subject treated for third molar surgery with piezoelectric surgery or rotating drills. The secondary outcomes chosen were changes in quality of life using a questionnaire form.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual wavelength low dose laser (Experimental): Immediately after suturing the patient, a low-dose laser application was performed on the laser group using the square probe (16 J/min) of the locally produced GRR laser device (Ankara, Turkey) for 5 minutes. The device combines a 22 mW GaAlAs infrared laser with a wavelength of 904 nm and a 10 mW red laser with a wavelength of 650 nm. The square probe contains 5 red lasers and 4 infrared lasers, covering an area of 30mm X 30mm.
  Interventions: Device: Dual wavelength low level laser
- Plasebo (Placebo Comparator): Laser probe will be applied to the control group patients, but the device was not operated.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Dual wavelength low level laser — Application of double wavelength low level laser to the related area after tooth extraction.
  Arms: Dual wavelength low dose laser
Device: Placebo — Only red light applied.
  Arms: Plasebo

SUMMARY:
Objective: To investigate the effects of single session dual wavelength low dose laser therapy to be applied after third molar tooth extraction on postoperative pain, edema and physical activities.

Materials and Methods: Thirty-six patients who applied for the extraction of a Class III and position B lower impacted wisdom tooth were included in the study. The patients were divided into 2 groups as laser and control group. Envelope selection method was used for randomization of patients. After the surgery, a single session of double wavelength low-dose laser therapy was applied to the patients. On the 2nd and 7th postoperative days, pain was measured with the VAS scale, edema was measured by face measurements of 3 different points, and quality of life was measured with the modified Posse scale.

DETAILED DESCRIPTION:
Objective and background: Pain, edema, and trismus are common problems after tooth extraction. Photobiomodulation therapy (PBMT) is frequently used as an adjunctive method to reduce these problems. However, there is no consensus in the literature regarding the type, power, session duration, and application frequency of the laser for this treatment method. The aim of this study is to examine the effectiveness of a single-session application of dual-wavelength PBMT (using a 904 nm GaAlAs infrared laser and a 650 nm red laser) on pain, edema, trismus, and the quality of life of patients following impacted mandibular third molar extraction.

Methods: The study included patients whose impacted mandibular third molars were to be extracted for prophylactic purposes. The patients were divided into two groups as the PBMT group and the placebo control group. Pain, swelling, maximum mouth opening, and quality of life parameters of the patients were evaluated.

ELIGIBILITY:
Inclusion Criteria:

ASA I 18-40 years aged

Exclusion Criteria:

Pregnancy Lactating, Anticoagulant or antiaggregant medication Radiotherapy to the head and face area, Allergy to local anesthetics and prescribed drugs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Swelling | Preoperative-Postoperative (Day 2 and 7)
  It was determined according to facial swelling measurements. Tragus and soft tissue pogonion, tragus and lateral corner of the mouth were measured and recorded with a flexible ruler.
Maximum Mouth Opening | Preoperative-Postoperative (Day 2 and 7)
  It is the procedure for determining the maximum mouth opening of the patient in mm. Measurements were determined as the distance between the incisal edges of the superior and inferior central teeth 11 and 41. In the absence of these teeth, other incisal teeth (21/31) in the adjacent half jaw were used. The maximum mouth opening determined before the operation was measured and recorded again on the 2nd and 7th days after the operation. The maximum mouth opening was measured with the help of a caliper.
Pain after surgery | Preoperative-Postoperative (Day 2 and 7)
  Pain assessment of the patient was done with visual analog scale (VAS). According to this evaluation, the line of a certain length was divided into 10 equal parts. 0 = no pain on the line, 5 = moderate pain, 10 = unbearable pain. This statement will also be verbally reported to the patient and the patient was asked to mark the severity of his pain on this hide.

SECONDARY OUTCOMES:
Operation Time | During the surgery
  The time from incision to the last suture was recorded.
Quality of Life of the Patients' | At 7th day.
  A questionnaire form evaluates quality of life. This questionnaire was divided into subscales corresponding to seven main adverse effects, and for each possible answer there was a score ranging from 0 to a variable number. It is a valid and reliable measure of the severity of symptoms after extraction of third molars, and of the impact of those symptoms on patients' perceived health.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farivar S, Malekshahabi T, Shiari R. Biological effects of low level laser therapy. J Lasers Med Sci. 2014 Spring;5(2):58-62. PMID 25653800
- [Background] Domah F, Shah R, Nurmatov UB, Tagiyeva N. The Use of Low-Level Laser Therapy to Reduce Postoperative Morbidity After Third Molar Surgery: A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2021 Feb;79(2):313.e1-313.e19. doi: 10.1016/j.joms.2020.09.018. Epub 2020 Sep 17. PMID 33058775